CLINICAL TRIAL: NCT02360774
Title: Mechanisms of Weight Loss With SGLT2 Inhibition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Jody Dushay, Principle Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014P000335
Record Dates: First submitted 2015-02-04; First posted 2015-02-11 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes; Overweight; Obesity
Keywords: Canagliflozin; Obesity; Weight Loss; Body Weight; Body Weight Changes; Overweight; Sodium-glucose transporter subtype 2 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Weight Loss; Body Weight; Body Weight Changes | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Canagliflozin (Experimental): Subjects will be randomized (1:1) to treatment with canagliflozin 300mg or placebo once daily for 18 weeks.
  Interventions: Drug: Canagliflozin
- Placebo (Placebo Comparator): Subjects will be randomized (1:1) to treatment with canagliflozin 300mg or placebo once daily for 18 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin — Subjects will take one 300mg capsule of canagliflozin or identically dispensed placebo by mouth once daily, for 18 weeks.
  Other Names: Invokana
  Arms: Canagliflozin
Drug: Placebo — Subjects will take one 300mg capsule of canagliflozin or identically dispensed placebo by mouth once daily, for 18 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of canagliflozin, a medication approved by the FDA for the treatment of type 2 diabetes, on body weight and metabolism in people with type 2 diabetes who are overweight or obese.

Canagliflozin lowers glucose levels in the blood by making the kidneys excrete, rather than absorb, glucose. Canagliflozin is also often associated with weight loss.

The study population will generally be type 2 diabetics, ages 18-75 years old, who are overweight or obese.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. BMI 25-45 kg/m2
3. Hemoglobin A1C > 6.5% but < 9%
4. Normal renal function (GFR > 60)
5. Age 18-75

Exclusion Criteria:

1. Type 1 diabetes
2. History of recurrent UTI or mycotic genital infections
3. Treatment with insulin or a GLP1 agent
4. Pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Canagliflozin: Subjects will take one 300mg capsule of canagliflozin once daily for 18 weeks.
- Placebo: Subjects will take one 300mg capsule of identically dispensed placebo by mouth once daily for 18 weeks.
Period: Overall Study
Arm/Group | Canagliflozin | Placebo
Started | 15 | 15
Completed | 12 | 13
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Canagliflozin | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants] — Population: 4 placebo dropouts, 2 treatment dropouts
  Participants
    number analyzed (Participants) | 12 | 13 | 25
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 12 | 13 | 25
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: dropouts
  years
    number analyzed (Participants) | 12 | 13 | 25
    (all) | 56.6 (1.98) | 61.8 (2.9) | 59.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: dropouts
  Participants
    number analyzed (Participants) | 12 | 13 | 25
    Female | 5 | 6 | 11
    Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: dropouts
  Participants
    number analyzed (Participants) | 12 | 13 | 25
    Hispanic or Latino | 1 | 1 | 2
    Not Hispanic or Latino | 11 | 12 | 23
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: dropouts
  Participants
    number analyzed (Participants) | 12 | 13 | 25
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 7 | 11
    White | 7 | 5 | 12
    More than one race | 1 | 1 | 2
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: dropouts
  participants
    United States: number analyzed (Participants) | 12 | 13 | 25
    United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Body weight will be measured at each study visit (screening visit, enrollment (study week 0), and at study weeks 2, 4, 8, 12 and 18). Change in body weight will be calculated using ANOVA such that body weight at all time points is included in the data analysis, rather than simply comparing weight at the enrollment visit to weight at the final study visit.
Time Frame: 18 weeks (duration of study)
Measure: Mean (Standard Error); unit: kg
Arm/Group | Canagliflozin | Placebo
Number analyzed (Participants) | 13 | 12
kg | 3.0 (0.7) | 0.3 (0.9)

2. Secondary Outcome: Change in Resting Energy Expenditure, Measured Using Indirect Calorimetery
Description: Resting energy expenditure will be measured at each study visit using indirect calorimetery. Data analysis will include change in REE from baseline to study conclusion, as well as change in REE throughout the study.
Time Frame: 18 weeks (duration of study)
Measure: Mean (Standard Error); unit: kcal
Arm/Group | Canagliflozin | Placebo
Number analyzed (Participants) | 13 | 12
kcal | -60.8 (54.4) | -68.6 (84.3)

3. Secondary Outcome: Change in Body Composition, Measured Using DXA Scanning.
Description: Body composition will be measured at baseline and at study completion using DXA scanning.
Time Frame: 18 weeks (duration of study)
Measure: Mean (Standard Error); unit: % fat
Arm/Group | Canagliflozin | Placebo
Number analyzed (Participants) | 13 | 12
% fat | -0.2 (0.4) | -0.4 (0.4)

4. Secondary Outcome: Change in Glycemic Control
Description: Hemoglobin A1C will be measured at baseline and at study completion.
Time Frame: 18 weeks (duration of study)
Measure: Mean (Standard Error); unit: percent glycated hemoglobin
Arm/Group | Canagliflozin | Placebo
Number analyzed (Participants) | 13 | 12
percent glycated hemoglobin | -0.4 (0.1) | -0.1 (0.2)

ADVERSE EVENTS:
Time Frame: duration of the study. each participant was enrolled for up to 18 weeks
Description: subjects were asked about AEs at each study visit
Arm/Group | Placebo | Canagliflozin
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/12 | 1/13
Other Adverse Events (participants affected / at risk) | 5/12 | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Canagliflozin (N=13)
pneumonia (Infections and infestations) | 0 (0) | 1 (1) — subject with known COPD experienced COPD flare and pneumonia requiring hospitalization.
infection (Infections and infestations) | 1 (1) | 0 (0) — subject experienced cellulitis following planned foot surgery
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — subject with known hepatic cyst had severe abdominal pain requiring hospitalization and drainage
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Canagliflozin (N=13)
hypoglycemia (Endocrine disorders) | 2 (2) | 2 (2) — blood sugar values < 70
polyuria (Renal and urinary disorders) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT02360774/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT02360774/Prot_SAP_001.pdf